CLINICAL TRIAL: NCT00779376
Title: Comparative, Randomized, Single-Dose, 2-Way Crossover Bioavailability Study of Ranbaxy and GlaxoSmithKline (Retrovir ® ) 300 mg Zidovudine Tablets in Healthy Adult Volunteers Under Fed Conditions
Brief Title: Bioequivalence Study of Zidovudine 300 mg Tablets, USP Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AA26101
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence
MeSH Terms: interventions — Zidovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Zidovudine 300mg tablets of Ranbaxy
  Interventions: Drug: Zidovudine 300mg tablets
- 2 (Active Comparator): Retrovir ®) 300 mg Zidovudine tablets of Glaxosmithkline
  Interventions: Drug: Zidovudine 300mg tablets

INTERVENTIONS:
Drug: Zidovudine 300mg tablets

SUMMARY:
The objective of this study was to assess the single-dose relative bioavailability of Ranbaxy and GlaxoSmithKline (Retrovir ®) 300 mg Zidovudine tablets, under fed conditions

DETAILED DESCRIPTION:
This was an open label, randomized, single dose, 2-way crossover, comparative bioavailability study performed on 68 healthy adult volunteers. In each period, subjects were housed from at least 10 hours before dosing until after the 12 hour blood draw. Single oral dose 300 mg Zidovudine doses were separated by a washout period of 7 days.

A total of sixty-eight (68) healthy adult subjects (29 males and 39 females) were enrolled in the study, of which sixty five (65) subjects (29 males and 36 females) completed the clinical portion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female volunteers, 18-55 years of age
2. Weighing at least 52 kg for males and 45 kg for females within 15 % of their ideal weights (table of 'Desirable weights of Adults', Metropolitan Life Insurance Company, 1983)
3. Medically healthy subjects with clinically normal laboratory profiles, vital signs and ECGs
4. Females of child bearing potential were either sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study or were using one of the following acceptable birth control methods:

   Surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) 6 months minimum; IUD in place for at least 3 months; Barrier methods (condom, diaphragm) with spermicide for at least 14 days prior to the first dose and throughout the study Surgical sterilization of the partner (vasectomy for 6 months minimum) Hormonal contraception for at least 3 months prior to the first dose of the study Other birth control method deemed acceptable
5. Postmenopausal women with amenorrhea for at least 2 years
6. Given voluntary written informed consent to participate in this study.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease
2. In addition history or presence of alcoholism or drug abuse within the past year, or hypersensitivity or idiosyncratic reaction to Zidovudine or to any other nucleoside analogue
3. Female subjects who were pregnant or lactating
4. Subjects who tested positive at screening for HIV, HBsAg or HCV
5. Subjects who have used any drugs or substances known to be strong inhibitors of cyp enzymes (formerly known as cytochrome p 450 enzymes) within 10 days prior to the first dose
6. Subjects who have used any drugs or substances known to be strong inducers of cyp enzymes (formerly known as cytochrome P 450 enzymes) within 28 days prior to the first dose and throughout the study
7. Subjects who through completion of the study would have donated in excess of 500 mL of blood in 14 days, 1500 mL of blood in 180 days or 2500 mL of blood in 1 year
8. Subjects who have participated in another clinical trial within 28 days prior to the first dose.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2005-02; Primary Completion 2005-03 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- MDS Pharma Services, Montreal, Quebec, Canada

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html